CLINICAL TRIAL: NCT01529333
Title: Middle Ear Implant With MET V for Mixed Hearing Loss
Brief Title: Middle-Ear Implant With MET V Transducer (Aka MET V System)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Otologics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G070237
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Mixed Conductive and Sensorineural Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Ossicular Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Middle Ear Implant with MET V Transducer — The MET V System is indicated for use in addressing the amplification needs of adults, 18 years of age and older, who have mixed hearing loss.

SUMMARY:
The purpose and objective of this study is to evaluate the safety and efficacy of the MET V System for the treatment of individuals with mixed hearing loss.

DETAILED DESCRIPTION:
The MET V System is an investigational, fully-implantable middle ear hearing prosthesis. A mixed hearing loss has both a sensorineural component and a conductive component that results when sound being delivered to an impaired cochlea is attenuated by a disordered outer or middle ear.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women, 18 years of age or older
* Moderate to severe mixed hearing loss, as a result of a combination of sensorineural hearing loss and chronic ear disease, prior failed tympanoplasties, severe otosclerosis, radical mastoidectomy, or congenital abnormality as evidenced by the following in the ear to be implanted:

  * Bone conduction thresholds are measurable at 0.5,1,2,3 and 4 kHz
  * Bone conduction thresholds are 20 dB or poorer at greater than 2 kHz
  * Air conduction thresholds are 35 dB or poorer at 0.5,1,2,3 and 4 kHz
* Air-bone gap in ear to be implanted is greater than 15 dB at three or more frequencies from 0.5 - 4 kHz
* Word recognition appropriate for sensorineural component of loss
* Non-fluctuating and stable hearing status

  a. as defined as by no significant change or progression in the bone conduction thresholds >15dB at two consecutive octaves for at least 12 months.
* English Speaking (fluent)
* Realistic expectations for the device
* Willingness to sign the informed consent and participate in the study

Exclusion Criteria:

* Vestibular disorder, including Meniere's Syndrome
* Recurring otitis media over the past year (>2/year)
* Non-organic hearing loss
* Retrocochlear hearing loss
* Central auditory nervous system disorder
* Medical contraindications to surgery or use of the device
* Women who are pregnant or at risk of becoming pregnant
* Developmentally delayed or manifesting organic brain dysfunction
* Persons with physical or geographic limitations that may render them incapable of completing scheduled study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
CNC Word Recognition Scores | Occurs at 3, 6, and 12 month follow-up visits
  * The primary efficacy endpoint is the mean change in the implant ear from CNC word recognition (unaided for mixed hearing loss and aided with hearing aid for sensorineural hearing loss) scores at the six month follow-up.
  * The secondary efficacy endpoints include a speech perception outcome (BKB-SIN) measure and a subjective questionnaire (APHAB). The endpoint for the BKB-SIN is the mean change in score at the six month follow-up compared to the control. The endpoint for the subjective questionnaire (APHAB)is post-operative responses compared to the pre-operative control responses.

SECONDARY OUTCOMES:
BKB-SIN and Subject Questionnaires | Will be monitored to 12 months
  * Primary safety endpoint is the mean change from baseline (average across 0.5, 1, 2, 3 4 kHz) in the implanted ear for pure tone bone conduction thresholds at the 6-month study visit, and safety will be monitored to 12 months.
  * Secondary safety endpoints include assessments of adverse events and device failures.